CLINICAL TRIAL: NCT02941679
Title: A 24-week, Randomized, Double-Blind, Active-controlled, Parallel Study of HCP1202 Combination Product, HGP1011, and HCP0910 in Treatment of Subjects With COPD
Brief Title: Clinical Efficacy and Safety Evaluation of HCP1202 in COPD Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-FLUT-301
Record Dates: First submitted 2016-10-14; First posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- HCP1202 (Experimental): Test
  Interventions: Drug: HCP1202
- HGP1011 (Active Comparator): Control
  Interventions: Drug: HGP1011
- HCP0910 (Active Comparator): Control
  Interventions: Drug: HCP0910

INTERVENTIONS:
Drug: HCP1202 — Hanmi Pharmaceutical. Co., Ltd.
  Other Names: HCP1202 Capsule
  Arms: HCP1202
Drug: HGP1011 — Boehringer Ingelheim
  Other Names: HGP1011 Capsule
  Arms: HGP1011
Drug: HCP0910 — GlaxoSmithKline
  Other Names: HCP0910 Capsule
  Arms: HCP0910

SUMMARY:
A phase 3 study to evaluate efficacy and safety of HCP1202

DETAILED DESCRIPTION:
This study is designed as a multi-center, double-blinded, randomized, phase 3 clinical trial to evaluate the efficacy and safety of HCP1202 compared to either treatment with HGP1011 or HCP0910 in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female adults aged ≥ 40 years.
* Patients diagnosed with COPD.
* Patients with FEV1/FVC < 0.7 at screening.
* Patients with a post-bronchodilator FEV1 < 60% of the predicted normal OR Patients with a post-bronchodilator FEV1 < 80% of the predicted normal if COPD exacerbation is moderate or worse developed at least twice within the past year or hospitalization occurred at least once within the past year due to COPD exacerbation.
* Patients with COPD Assessment Test ≥ 10.
* Patients with a history (current or ex-smokers) of smoking 10 pack-years or more (e.g. 10 pack years = 1 pack/day x 10 years, or ½ pack/day x 20 years).
* Patients who understand the process of clinical trial and signed written informed consent.

Exclusion Criteria:

* Patients with a current diagnosis of asthma.
* Patients with the following lung disorders that can affect the clinical trial, except for COPD: lung cancer, interstitial lung disease, thromboembolic pulmonary disease, moderate to severe bronchiectasis, sarcoidosis, pulmonary fibrosis, pulmonary hypertension, active tuberculosis, clinically significant tuberculous destroyed lung, alpha1-antitrypsin deficiency, etc.
* Patients underwent pulmonary lobectomy or lung volume reduction surgery within the past year.
* Patients who developed COPD exacerbation where antibiotics and/or systemic corticosteroids and/or hospitalization is advisable within 4 weeks prior to Visit 1 or during Run-in period (but, re-screening is possible 4 weeks after resolution of the COPD exacerbation occurred within 4 weeks prior to Visit 1).
* Patients who administered antibiotics for lower respiratory infection within 4 weeks prior to Visit 1 or during Run-in period (but, re-screening is possible 4 weeks after resolution of COPD exacerbation occurred within 4 weeks prior to Visit 1).
* Patients who have changed the COPD treatment method within 12 weeks prior to Visit 1 (but, PDE4 inhibitor can be used until 4 weeks prior to Visit 1).
* Patients administered systemic corticosteroids within 4 weeks prior to Visit 1.
* Patients with the following clinically significant cardiovascular diseases: a history of myocardial infarction or unstable angina within 6 months prior to Visit 1, a history of unstable arrhythmia where its therapy method has been changed within 1 year prior to Visit 1, a history of hospitalization from NYHA Class III-IV heart failure, a history of atrial fibrillation, negative cardiac tachycardia, and/or hypertrophic cardiomyopathy.
* Patients with a history of long QTc syndrome.
* Patients with the clinical significance of ECG abnormality at screening (QTc(F) ≥ 470 ms).
* Patients who require long-term oxygen therapy for more than 12 hours a day.
* Patients participated in acute respiratory rehabilitation within 6 months prior to Visit 1 (except for the patients under stabilized respiratory rehabilitation therapy of at least 6 weeks).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-02 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Trough FEV1 at Week 12 | Baseline, Week 12

SECONDARY OUTCOMES:
Change from Baseline in Trough FEV1 at Week 4 & 8 | Baseline, Week 4, Week 8
Change from Baseline in Trough FVC at Week 4 & 8 & 12 | Baseline, Week 4, Week 8, Week 12
Change from Baseline in Trough FEV1/FVC at Week 4 & 8 & 12 | Baseline, Week 4, Week 8, Week 12
Transition Dyspnea Index scores at Week 4 & 8 & 12 | Week 4, Week 8, Week 12
Change from Baseline in Total SGRQ-C (St. George's Respiratory Questionnaire for COPD patients) and sectional scores at Week 4 & 8 & 12 | Baseline, Week 4, Week 8, Week 12
Percentage (%) of Subjects Experienced with Moderate to Severe COPD Exacerbation from Baseline to Week 12 | Baseline through Week 12
Number of Occurrences in Moderate to Severe COPD Exacerbation per Subject from Baseline to Week 12 | Baseline through Week 12
Total Amount of Rescue Medication Used per Subject from Baseline to Week 12 | Baseline through Week 12
Average Daily Use of Rescue Medication per Subject from Baseline to Week 12 | Baseline through Week 12

CONTACTS AND LOCATIONS:
Overall Officials: HyoungKyu Yoon, M.D., Ph.D., Principal Investigator — Yeouido St. Mary's Hospital

IPD SHARING:
Plan to Share IPD: No